CLINICAL TRIAL: NCT01267123
Title: The Value of the Trendelenburg Position During Routine Colonoscopy: A Pilot Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1173017
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Colonoscopy
MeSH Terms: interventions — Head-Down Tilt; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trendelenburg position (Experimental): The endoscopist places the patient in 15° Trendelenberg position immediately prior to the initiation of the colonoscopy.
  Interventions: Procedure: Trendelenburg position
- Standard care (Other): The patient will have colonoscopy in the standard horizontal position
  Interventions: Procedure: Standard care

INTERVENTIONS:
Procedure: Trendelenburg position — The patient will be placed in the Trendelenburg position with a 15 degree angle of inclination
  Other Names: Head-Down Tilt
  Arms: Trendelenburg position
Procedure: Standard care — The patient will be placed in the standard horizontal position
  Arms: Standard care

SUMMARY:
Colonoscopy is a procedure commonly performed to screen for colon cancer and to look for and remove colon polyps. It involves inserting a flexible tube, equipped with a video-camera at the tip, through the colon. The insertion process can be difficult in some patients, resulting in an uncomfortable and lengthy procedure.We postulate that raising the foot of the bed so that the stretcher forms a 15 degrees angle with the floor ("Trendelenburg position") may make the colonoscopy easier and more comfortable to the patient.

DETAILED DESCRIPTION:
Colonoscopy is a procedure commonly performed to screen for colon cancer and to look for and remove colon polyps. It involves inserting a flexible tube, equipped with a video-camera at the tip, through the colon. The insertion process can be difficult in some patients, resulting in an uncomfortable and lengthy procedure. Colonoscopy procedures are typically started with the patient positioned on their left side. If there is later difficulty advancing the colonoscope, the patient is shifted to other positions (e.g. back, right side, prone). We postulate that raising the foot of the bed so that the stretcher forms a 15 degrees angle with the floor ("Trendelenburg position") may make the colonoscopy easier and more comfortable to the patient. This is a position commonly used in gynecologic surgery. This is a pilot project for us to gain experience with doing colonoscopy this way. The enrolled patient will be assigned randomly to 2 groups: one in the standard left lateral position and one in the 15 degree Trendelenberg position. We will be collecting data regarding the procedure from each group in the form of questionnaire and data sheet which will be filled during or at the conclusion of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient age between 18-75 years old.
* Colonoscopy performed for polyp surveillance or colon cancer screening purposes.
* Patient able to provide informed consent.

Exclusion Criteria:

* History of colon resection
* History of inflammatory bowel disease
* Pregnancy
* History of ischemic optic neuropathy or glaucoma
* Patient unable to provide informed consent
* Patients who did not fast for ≥2 hours prior to presenting for the procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The time of the procedure from the insertion of the colonoscope until the cecal base is reached | This outcome is measured when the cecum is intubated during a colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Abdo M Saad, MD, Principal Investigator — University of Missouri-Columbia

IPD SHARING:
Plan to Share IPD: Undecided